CLINICAL TRIAL: NCT03363269
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Evaluate the Efficacy and Safety of ID1201 for Dose-finding in Mild Alzheimer's Disease
Brief Title: Evaluate the Efficacy and Safety of ID1201 for Dose-finding in Mild Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID-BOA-201
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ID1201 100mg (Experimental)
  Interventions: Drug: ID1201
- ID1201 200mg (Experimental)
  Interventions: Drug: ID1201
- ID1201 400mg (Experimental)
  Interventions: Drug: ID1201
- Placebo (Placebo Comparator)
  Interventions: Drug: ID1201

INTERVENTIONS:
Drug: ID1201

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of ID1201 in patients with mild Alzheimer's disease

DETAILED DESCRIPTION:
ID1201 is a fruit extract of Melia toosendan. ID1201 alleviates Alzheimer's disease-type pathologies and cognitive deficit through the various actions of its effective components such as α-secretase activation followed to Aβ reduction, RAGE inhibition, neuro-protection, and anti-inflammatory activities.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with dementia of Alzheimer's type according to DSM-IV criteria and probable Alzheimer's disease according to the NINCDS-ADRDA
2. modified Hachinski Ischemia Scale score of less than or equal to 4
3. Mini-Mental State Examination score 16 to 26 and Clinical Dementia Rating-Global Scale score 0.5 to 1
4. Amyloid postivie PET image (BAPL score 2 or 3)
5. Patients who have not received AChE inhibitors or NMDA antagonist at least for 3 months prior to the screening visit

Exclusion Criteria:

1. Patients diagnosed or accompanied with Dementia due to other Neurodegenerative disorders other than Alzheimer's disease
2. Chronic alcohol and/or drug abuse within the past 5 years
3. Subjects who have medical history of significant renal disease (ccr<30ml/min) or hepatic disease( 3*ULN <= ALT or AST)
4. Has received choline agonists, anticholinergics, anticonvulsants, antidepressants, antipsychotic drugs, Ginko biloba extract, Vitamin E, hormone replacement therapy etc. in the previous 4 weeks

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog11) at 12 Weeks | Baseline, 12 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- South Korea (20):
  - Dong-A University Hospital, Busan
  - Changwon Fatima Hospital, Changwon
  - Kangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Myongji Hospital, Goyang
  - Hanyang University Guri Hospital, Guri-si
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Bundang Hospital, Seongnam-si
  - Chung-Ang University Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - KunKuk University Hospital, Seoul
  - Ajou University Medical Center, Suwon
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No